CLINICAL TRIAL: NCT06288438
Title: Multicomponent Telerehabilitation to Engage Veterans in Effective Self-Management of ComplexHealth Conditions
Brief Title: Multicomponent Telerehabilitation to Engage Veterans in Effective Self-Management of Complex Health Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E5012-R; 23-2306 (Other: COMIRB)
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Multimorbidity; Physical Deconditioning
Keywords: telerehabilitation; high intensity; biobehavioral; social support; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 2 groups. Group 1 will receive the intervention for 24 weeks. Group 2 will receive the control condition for 24 weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multicomponent Telerehabilitation Intervention (Group 1) (Experimental): Veterans randomized to the MCTR group will complete the 24-week study intervention consisting of the Active (weeks 1-6), Transition (weeks 7-12), and Sustainability (weeks 13-24) phases. Participants will receive a total of 16 individual sessions (6 integrated, 4 high-intensity rehabilitation, and 6 self-management intervention sessions).
  Interventions: Behavioral: Motivational Interviewing Techniques; Other: Physical Therapy Interventions
- Education Control (Group 2) (Other): This group will not receive any exercise intervention but will complete 16 sessions with research staff through videoconferencing. These visits will consist of standardized Health Status Update and education sessions on general health topics.
  Interventions: Other: Education; Other: Health Status Updates; Other: Physical Therapy Consult

INTERVENTIONS:
Behavioral: Motivational Interviewing Techniques — Motivational Interviewing Techniques including but not limited to open-ended questions, reflection, affirmations, and summary will be used to build participant rapport, support behavior change (physical activity), and facilitate program engagement.
  Arms: Multicomponent Telerehabilitation Intervention (Group 1)
Other: Physical Therapy Interventions — Strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise.
  Arms: Multicomponent Telerehabilitation Intervention (Group 1)
Other: Education — Education on general health topics which may include the following: basic nutrition, stress reduction, sleep hygiene, etc.
  Arms: Education Control (Group 2)
Other: Health Status Updates — Health Status Updates will be completed by a trained assessor. The assessor will ask about adverse events, general health topics, medication changes, and changes in social circumstances.
  Arms: Education Control (Group 2)
Other: Physical Therapy Consult — Participants in the control condition will be offered a physical therapy consult at the end of their 24 week study involvement.
  Arms: Education Control (Group 2)

SUMMARY:
Medically complex older Veterans are at greater risk for progressive declines in physical function, lower quality of life, and increasing care needs. Additionally, older Veterans experience social isolation and loneliness, and have low levels of physical activity. While the Veterans Health Administration has established programs to address rehabilitation needs, these programs tend to be diagnosis-focused, lack self-management approaches, include low-intensity rehabilitation, and typically require in-person attendance. A MultiComponent TeleRehabilitation (MCTR) program that includes high-intensity rehabilitation and self-management interventions, social support, and telehealth and technology supports may be more effective in improving and sustaining physical function for older Veterans with complex health conditions. Therefore, this project is designed to determine whether the MCTR program improves strength and physical function more effectively than traditional interventions.

DETAILED DESCRIPTION:
The proposed MultiComponent TeleRehabilitation (MCTR) program addresses current healthcare deficiencies by using a multicomponent approach that includes both high-intensity rehabilitation interventions and self-management interventions that are not part of traditional physical therapy interventions. Therefore, the investigators propose a two-arm, parallel randomized trial using a crossover study design to determine the effectiveness (AIM 1) of a 12-week multicomponent telerehabilitation program to improve physical function. The investigators will also measure Veterans' clinical outcomes to evaluate the effectiveness of the MCTR program to improve physical activity, health self-management, and self-reported health (AIM 2). Lastly, the investigators will explore the effects of the MCTR program on safety events such as emergency room visits, hospitalizations, falls, and other adverse events (AIM 3). Participants (n=126) will be randomized to MCTR or Control group using computer-generated random blocks, stratified by sex. The MCTR group will participate in the 24-week program consisting of 1) progressive, high-intensity rehabilitation, 2) self-management interventions, 3) social support, and 4) technology supports. The 12-week program is split into three phases: the Active Phase (weeks 1-6), the Transition Phase (weeks 7-12), and the Sustainability Phase (weeks 13-24). The Control group will participate in education and health status update sessions in parallel to the MCTR 12-week program. Outcomes will be collected at baseline, 6 weeks, 12 weeks (primary endpoint), and 24 weeks. Achievement of the proposed aims will provide evidence to expand high quality telerehabilitation services for medically complex older Veterans with multiple factors contributing to poor health (e.g., social isolation, loneliness, physical inactivity, poor self-management). Importantly, results will guide the advancement of rehabilitation practices, moving away from a traditionally narrow, episodic, diagnosis-focused approach to a model emphasizing whole health self-management and sustained healthy living. Study findings will have immediate clinical impact as they will be directly translatable to other medically complex and underserved populations who will benefit from innovative telerehabilitation care approaches.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and older
* Multiple chronic conditions (Functional Comorbidity Index > or = 3)
* Impaired physical function (< or = 8 repetitions on 30 second sit to stand test)

Exclusion Criteria:

* Life expectancy < 12 months
* Acute or progressive neurological disorder (e.g. amyotrophic lateral sclerosis, recent stroke)
* Moderate to severe dementia (<11 on telephone Montreal Cognitive Assessment(T-MoCA))
* Medical conditions precluding safe participation in high-intensity rehabilitation (e.g. unstable angina)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
2 Minute Step Test | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This is a functional performance test for aerobic endurance. It requires participants to march in place for 2 minutes (alternating legs), and the score is the number of repetitions completed on the right leg. Scores are continuous, and higher scores indicate better aerobic endurance.

SECONDARY OUTCOMES:
Arm Curl Test | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This is a functional performance test for upper body strength and is performed on each arm (one arm at a time). It requires the participant to perform as many arm curls (biceps curls) as possible in 30 seconds. Males use a 8 pound weight and females use a 5 pound weight. Scores are continuous, and higher scores indicate greater arm strength (better outcome)
30 Second Sit To Stand | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  The test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More repetitions indicate better lower extremity strength.
Physical Activity | Will be collected at Baseline, 12 weeks, and 24 weeks.
  Physical activity will be measured via accelerometry and will include an averaged daily step count.
Exercise readiness to change | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  Four-item survey collected via interview format, and it is used to categorize participants into stages of change according to the Transtheoretical Model, possible stages include: (pre-contemplating, contemplation, preparation, action, and maintenance).
Self-efficacy for Exercise Scale | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  A 9-item survey, each item is scored on a scale of 0 (not confident) to 10 (very confident) and higher scores indicate greater self-efficacy.
Self-efficacy of Managing Chronic Conditions | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  A 8-item survey rated on a 5-point Likert scale [I am not at all confident (1) to I am very confident (5)], and higher scored indicates better self-efficacy.
The Patient-Specific Functional Scale | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This is a questionnaire collected via interview format that quantifies activity or participation limitations that are important to the patient. Each participant identifies 3 activities that are important and that they are currently unable to do or having difficult performing due to their health; each item is then rated on a 0 (unable to preform activity) 0 to 10 (able to perform activity at the same level as before injury or problem) scale. The total score is an average of the 3 activities.
Activity Measure for Post-Acute Care (AM-PAC) basic mobility outpatient routine short form | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This questionnaire consists of 18 items rated on a 4-point Likert scale in response to the prompt, "How much difficulty do you currently have..." Total scores range from 18 to 72 and higher scores indicate less difficulty with physical tasks.
Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 (PROPr) survey | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This is a 29-item questionnaire, and most items are rated on a 5-point Likert scale. There is one pain intensity item rated on a 0 (no pain) to 10 (worst pain imaginable) scale. Higher scores indicate more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) v2 social isolation short form (SF) 8a | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  An 8-item questionnaire rated on a 1 (never) to 5 (always) Likert scale. Higher scores indicate greater perceptions of loneliness and isolation, which is considered a worse outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) satisfaction with participation in discretionary social activities short form (SF) 7a | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  Includes 7 items rated on a 1 (not at all) to 5 (very much) Likert scale. Higher scores indicate greater satisfaction with discretionary social activities.
Physical Activity and Social Support Scale | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  A 20 -item survey rated on a scale of 1 (never true) to 7 (always true) that measures emotional, informational, instrumental, validation, and companionship support related to physical activity. Higher scores indicated greater levels of perceived social support.
Geriatric Pain Measure | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  Consists of 22 items scored as yes (1 point) or no (0 points) that assess whether or not a person does or would have pain during activities. There are also 2 items measured on a scale of 0 (no pain) to 10 (worst pain). Total scores range from 0-42 and adjusted scores range from 0-100 with higher scores indicating worse pain.
Pain Coping Inventory | Change from baseline to 6 weeks, 12 weeks, and 24 weeks compared to the control group.
  This measures both active (transformation, distraction, reducing demands) and passive (retreating, worrying, resting) coping strategies. The inventory includes 34 items rated on a scale from 1 (hardly ever) to 4 (very often). Higher scores indicate more frequent use of each specific coping strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No